CLINICAL TRIAL: NCT05100667
Title: A Potential Role for Oxygen in the Development of Mental Fatigue and the Subsequent Decline in Cognitive Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principal investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 796
Record Dates: First submitted 2021-01-28; First posted 2021-10-29 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Mental Fatigue; Near Infrared Spectroscopy; NIRS; Hypoxia; Cerebral Heamodynamics; Cognition
MeSH Terms: conditions — Mental Fatigue; Hypoxia

STUDY DESIGN:
Intervention Model Description: randomized blinded placebo-controlled counterbalanced crossover design
Who Masked: Participant
Masking Description: We will inform the participants in a way that explains the study as an investigation about the influence of different cognitive tasks on a subsequent physical task at various altitudes looking at other physiological outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental fatigue (Experimental): Stroop task
  Interventions: Other: Hypoxia; Other: Normoxia
- Control MF (Placebo Comparator): Emotionally neutral documentary
  Interventions: Other: Hypoxia; Other: Normoxia

INTERVENTIONS:
Other: Hypoxia — altitude (3800m)
  Other Names: Mental fatigue
Other: Normoxia — sea level
  Other Names: Mental fatigue

SUMMARY:
Introduction Both Mental Fatigue (MF) and hypoxia impair multiple aspects of cognitive functioning. The decline in cognitive functioning in hypoxic conditions is associated with alterations in brain oxygenation and hemodynamic responses. These hemodynamic responses are preferably measured at the prefrontal cortex, an area of the brain that is known for its executive function and role in decision making, planning, attention and (short-term) memory. This study will investigate the role of prefrontal cortex oxygenation during the development of mental fatigue and during cognitive performances by altering the ambient oxygen availability through normobaric hypoxia (3800m; 12,9% O2) and normoxia.

Methods Subjects will perform four trials in a sound-insulated climate chamber (20°C and 40% RH). Upon entry in the climatic chamber participants will adapt to the environment for 30 minutes. Next, they will perform a modified cognitive test battery "cognition", a fine motor task "Motor Performance Series" and a visuomotor-fitlight task before and after a 60-minute individualized Stroop task or control task (randomized. blinded, placebo controlled, counter-balanced, cross-over design). Nearinfrared spectroscopy (NIRS) will be used to assess hemodynamic changes (oxygenated hemoglobin (O2Hb), deoxygenated-hemoglobin (HHb) and total hemoglobin (tHb)) at the PFC.

Hypotheses 1) MF will lead to earlier changes in the prefrontal NIRS-parameters (O2Hb, HHb, tHb) with lower oxygen availability. 2) The effects of MF on cognitive performance manifest itself to a greater extent with lower oxygen availability.3) Visuomotor performance declines to a greater extent due to MF with lower oxygen availability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological or cardiovascular disorders)
* Male or female
* No medication
* Non-smoker
* Between 18 and 35 years old
* Recreational athlete population; performance level 2 or 3 for men according to De Pauw et al. (2013)[29] and performance level 2 or 3 for woman according to Decroix et al. (2015)
* Non-acclimatized to altitude (at least 2 months)

Exclusion Criteria:

* Injuries
* Acclimated to altitude
* Use of medication
* Use of caffeine and heavy efforts 24 hours prior each trial
* Not eating a standardized meal, the morning of each trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral oxygenation | 2 hours
  Prefrontal cortex oxygenation = relative changes in oxy- and deoxy hemoglobin at the prefrontal cortex. During the whole frame, participants are equipped with a Near Infrared Spectroscopy device that measures cerebral oxygenation continuously at 10hz.
Mental fatigue | 60 minutes
  Results of a visual analogue scale for mental fatigue

SECONDARY OUTCOMES:
Cognition | 20 minutes
  Results of the Joggle cognition test battery (accuracy and reaction time
Fine motor control | 5 minutes
  Results of the vienna test system (MLS) =accuraccy and reaction time
Visuomotor control | 7 minutes
  Results of a visuomotor fitlight task = accuracy and reaction time

OTHER OUTCOMES:
Hemoglobin concentration | 10 minutes
  Hemoglobin will be assessed through the analysys of 1 drop of arterial blood
Blood glucose concentration | 10 minutes
  Hemoglobin will be assessed through the analysys of 1 drop of arterial blood

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Human Physiology - MFYS, Brussels, Brussels Capital
  - Human Physiology - MFYS, Brussels

IPD SHARING:
Plan to Share IPD: Undecided